CLINICAL TRIAL: NCT02556450
Title: Bioprofiling Response to Mineralocorticoid Receptor Antagonists for the Prevention of Heart Failure. A Proof of Concept Clinical Trial Within the EU FP 7 (European Union FP7) "HOMAGE" Programme " Heart OMics in AGing "
Brief Title: Bioprofiling Response to Mineralocorticoid Receptor Antagonists for the Prevention of Heart Failure
Acronym: Homage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ACS Biomarker (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Homage
Record Dates: First submitted 2015-09-08; First posted 2015-09-22 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spironolacton Group (Experimental): Spironolacton Sandoz given 25mg daily oral use
  Interventions: Drug: Spironolacton
- Control group (No Intervention): Only background treatment

INTERVENTIONS:
Drug: Spironolacton — Administration of Spironolacton 25 mg per day
  Other Names: Spironolacton Sandoz
  Arms: Spironolacton Group

SUMMARY:
Despite advances in care, prognosis remains poor once overt Heart Failure (HF) has developed. Prevention is most efficient when directed toward patients at risk and when mechanistically targeted to patients most likely to respond. An increase in myocardial and possibly vascular collagen content (fibrosis) may be a major determinant of the transition to HF. In patients with hypertension and diabetes, two important risk-factors for HF, changes in blood markers of fibrosis occur before clinically overt HF develops. These markers are also related to prognosis.

In the general population, Galectin-3 (Gal-3), a potential marker of fibrosis, is associated with cardiovascular (CV) risk factors, and predicts development of HF. In animal models, Gal-3 is a key mediator of aldosterone-induced CV and renal fibrosis and dysfunction.

The investigators hypothesize that the mineralocorticoid receptor antagonist (MRA), spironolactone, may prevent HF by acting on extracellular matrix remodelling, especially in patients with active fibrogenesis, identified by high Gal-3 levels. The benefit/risk ratio of spironolactone might be superior in patients with a higher compared to lower plasma concentrations of Gal-3.

Main objective is to investigate whether spironolactone can favourably alter extra-cellular matrix remodelling, assessed by changes in the fibrosis biomarker Procollagen Type III N-Terminal Peptide (PIIINP), in patients at increased risk of developing heart failure and whether this effect is greater in patients with increased plasma concentrations of Gal-3.

DETAILED DESCRIPTION:
The investigators hypothesize that the mineralocorticoid receptor antagonist (MRA), spironolactone, may prevent HF by acting on extracellular matrix remodelling, especially in patients with active fibrogenesis, identified by high Gal-3 levels. The benefit/risk ratio of spironolactone might be superior in patients with a higher compared to lower plasma concentrations of Gal-3.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent will be obtained prior to any study procedure;
* Age >60 years
* Clinical risk factors for developing heart failure, either:

  1. Coronary artery disease (h/o myocardial infarction, angioplasty or coronary artery bypass) Or
  2. At least two of the following:

     * Diabetes Mellitus requiring Hypoglycaemic Pharmacotherapy
     * Receiving pharmacological treatment for Hypertension
     * Microalbuminuria
     * Abnormal ECG (left ventricular hypertrophy, QRS >120msec, abnormal Q-waves)
* Biological risk: NT-pro-BNP values between 125 and 1,000 ng/L or BNP values between 35 and 280 pg/ml (consistent with ESC guidelines indicating risk of HF but helping to rule out prevalent HF or atrial fibrillation which are associated with marked increases in NT-proBNP/BNP and should be investigated)

Exclusion Criteria:

* Recent wound healing/inflammation:
* Surgical procedure, coronary, cerebral or peripheral vascular events or infection in the prior 3 months
* Cancer
* Autoimmune disease
* Hepatic Disease
* Pre-existing diagnosis of clinical HF
* Moderate/severe LV systolic ventricular dysfunction, i.e. LVEF <45%
* Moderate or severe valve disease (investigators opinion)
* eGFR< 30ml/min
* Serum potassium >5.0 mmol/L
* Treatment with an MRA or a loop diuretic (furosemide, bumetanide, ethacrynic acid or torasemide) in the previous three months
* Potassium supplements or potassium-sparing diuretic at time of enrolment.
* Atrial fibrillation within one month prior to inclusion (AF lasting <60 seconds on ambulatory ECG monitoring is permitted)

  •. History of hypersensitivity to spironolactone.
* Requiring treatment with prohibited medication according to SmPC with exception of ACE inhibitors or angiotensin receptor blockers
* Patients unable to give written informed consent.
* Participation in another interventional trial in the preceding month
* Ability to walk is, in the investigators opinion, clearly limited by joint disease or other locomotor problems rather than by cardiorespiratory fitness

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2016-01; Primary Completion 2018-09-30 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in serum concentrations of PIIINP | 9 months
  mmol/l

SECONDARY OUTCOMES:
changes in serum plasma levels of Biomarkers | 9 months
  PICP (synthesis), ICTP (degradation) and GAL3
Cardiac remodelling 1 | 9 months
  NT-proBNP (ELISA, central Lab), from baseline to 9 months (Certified centers and central readings).
Cardiac remodelling 2 | 9 months
  Left Ventricular Mass (g/m)
Cardiac remodelling 3 | 9 months
  Left Atrial Volume (ml)
Cardiorespiratory performance during exercise | baseline, 9 months
  Shuttle walk test: Distance walked in meters
Vascular function | screening, baseline, month1, month3, month 6, month 9
  non-invasive technologies: BP lab Audicor system
heart failure or AF | 9 months
  Rate of the clinical composite of development of heart failure or atrial fibrillation, non-fatal myocardial infarction or stroke or CV death from baseline to 9 months. The HOMAGE blinded clinical event committee will adjudicate all serious adverse events.
Adverse events | screening, baseline, month1, month3, month 6, month 9
  All adverse events
Worsening renal function | screening, baseline, month1, month3, month 6, month 9
  decline in eGFR >20%
Hyperkalemia | screening, baseline, month1, month3, month 6, month 9
  rise of serum potassium to >5.5 mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: John Cleland, PhD, Principal Investigator — Imperial College London
Locations (9):
- France (2):
  - Hopital Sud Francilien, Corbeil-Essonnes
  - CHU de Nancy, Nancy
- Charite Universitatsmedizin Berlin, Kardiologie, Berlin, Germany
- St, Michaels Hospital, Dublin, Ireland
- Santa Margherita Hospital, Cortona, Italy
- Maastricht University Medical Center, Maastricht, Netherlands
- United Kingdom (3):
  - Queen Elizabeth University Hospital, Glasgow
  - Castle Hill Hospital, Hull
  - Central Manchester University Hospitals NHS, Manchester

REFERENCES:
- [Derived] Yu YL, Siwy J, An DW, Gonzalez A, Hansen T, Latosinska A, Pellicori P, Ravassa S, Mariottoni B, Verdonschot JA, Ahmed F, Petutschnigg J, Rossignol P, Heymans S, Cuthbert JJ, Girerd N, Clark AL, Verhamme P, Nawrot TS, Janssens S, Cleland JG, Zannad F, Diez J, Mischak H, Ferreira JP, Staessen JA; HOMAGE investigators. Urinary proteomic signature of mineralocorticoid receptor antagonism by spironolactone: evidence from the HOMAGE trial. Heart. 2024 Sep 16;110(19):1180-1187. doi: 10.1136/heartjnl-2023-323796. PMID 38729636
- [Derived] Monzo L, Ferreira JP, Cleland JGF, Pellicori P, Mariottoni B, Verdonschot JAJ, Hazebroek MR, Collier TJ, Cuthbert JJ, Pieske B, Edelmann F, Petutschnigg J, Khan J, Ahmed FZ, Girerd N, Bozec E, Diez J, Gonzalez A, Clark AL, Cosmi F, Staessen JA, Heymans S, Rossignol P, Zannad F. Dyskalemia in people at increased risk for heart failure: findings from the heart 'OMics' in AGEing (HOMAGE) trial. ESC Heart Fail. 2022 Dec;9(6):4352-4357. doi: 10.1002/ehf2.14086. Epub 2022 Sep 6. PMID 36065795
- [Derived] Verdonschot JAJ, Ferreira JP, Pizard A, Pellicori P, Brunner La Rocca HP, Clark AL, Cosmi F, Cuthbert J, Girerd N, Waring OJ, Henkens MHTM, Mariottoni B, Petutschnigg J, Rossignol P, Hazebroek MR, Cleland JGF, Zannad F, Heymans SRB; HOMAGE "Heart Omics in AGEing" Consortium. The Effect of Spironolactone in Patients With Obesity at Risk for Heart Failure: Proteomic Insights from the HOMAGE Trial. J Card Fail. 2022 May;28(5):778-786. doi: 10.1016/j.cardfail.2021.12.005. Epub 2021 Dec 18. PMID 34933097
- [Derived] Verdonschot JAJ, Ferreira JP, Pellicori P, Brunner-La Rocca HP, Clark AL, Cosmi F, Cuthbert J, Girerd N, Mariottoni B, Petutschnigg J, Rossignol P, Cleland JGF, Zannad F, Heymans SRB; HOMAGE "Heart Omics in AGEing" consortium. Proteomic mechanistic profile of patients with diabetes at risk of developing heart failure: insights from the HOMAGE trial. Cardiovasc Diabetol. 2021 Aug 9;20(1):163. doi: 10.1186/s12933-021-01357-9. PMID 34372849
- [Derived] Ferreira JP, Verdonschot J, Wang P, Pizard A, Collier T, Ahmed FZ, Brunner-La-Rocca HP, Clark AL, Cosmi F, Cuthbert J, Diez J, Edelmann F, Girerd N, Gonzalez A, Grojean S, Hazebroek M, Khan J, Latini R, Mamas MA, Mariottoni B, Mujaj B, Pellicori P, Petutschnigg J, Pieske B, Rossignol P, Rouet P, Staessen JA, Cleland JGF, Heymans S, Zannad F; HOMAGE (Heart Omics in AGEing) Consortium. Proteomic and Mechanistic Analysis of Spironolactone in Patients at Risk for HF. JACC Heart Fail. 2021 Apr;9(4):268-277. doi: 10.1016/j.jchf.2020.11.010. Epub 2021 Feb 3. PMID 33549556
- [Derived] Pellicori P, Ferreira JP, Mariottoni B, Brunner-La Rocca HP, Ahmed FZ, Verdonschot J, Collier T, Cuthbert JJ, Petutschnigg J, Mujaj B, Girerd N, Gonzalez A, Clark AL, Cosmi F, Staessen JA, Heymans S, Latini R, Rossignol P, Zannad F, Cleland JGF. Effects of spironolactone on serum markers of fibrosis in people at high risk of developing heart failure: rationale, design and baseline characteristics of a proof-of-concept, randomised, precision-medicine, prevention trial. The Heart OMics in AGing (HOMAGE) trial. Eur J Heart Fail. 2020 Sep;22(9):1711-1723. doi: 10.1002/ejhf.1716. Epub 2020 Jan 16. PMID 31950604
- [Derived] Ferreira JP, Verdonschot J, Collier T, Wang P, Pizard A, Bar C, Bjorkman J, Boccanelli A, Butler J, Clark A, Cleland JG, Delles C, Diez J, Girerd N, Gonzalez A, Hazebroek M, Huby AC, Jukema W, Latini R, Leenders J, Levy D, Mebazaa A, Mischak H, Pinet F, Rossignol P, Sattar N, Sever P, Staessen JA, Thum T, Vodovar N, Zhang ZY, Heymans S, Zannad F. Proteomic Bioprofiles and Mechanistic Pathways of Progression to Heart Failure. Circ Heart Fail. 2019 May;12(5):e005897. doi: 10.1161/CIRCHEARTFAILURE.118.005897. PMID 31104495

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT02556450/SAP_000.pdf